CLINICAL TRIAL: NCT03550651
Title: Evaluation Of Antiplaque Efficacy Of Licorice Extract Mouthrinse & Hypertonic Salt Solution And Their Comparison With Essential Oil & Chlorhexidine Mouthrinses-An Invitro & Invivo Study"
Brief Title: Evaluation of Antiplaque Efficacy of Licorice Extract Mouthrinse & HSS and Their Comparison With EO & CHX Mouthrinse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government College of Dentistry, Indore (Other)
Responsible Party: Principal Investigator, Dr. Ruchi Gulati, Post Graduate Student, Government College of Dentistry, Indore
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: RGulati
Record Dates: First submitted 2018-03-10; First posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Mild Gingivitis; Periodontal Diseases; Plaque
Keywords: Plaque; Plaque regrowth; Licorice extract; Mouthrinse; Chlorhexidine mouthrinse; Hypertonic salt solution; Essential oils
MeSH Terms: conditions — Periodontal Diseases; Plaque, Amyloid | interventions — Glycyrrhiza glabra extract; Oils, Volatile; chlorhexidine gluconate; Chlorhexidine

STUDY DESIGN:
Intervention Model Description: 5x5 latin cross over study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Licorice extract mouthrinse (Experimental): 10ml twice a day for 4 Days.
  Interventions: Other: Licorice
- Hypertonic salt solution (Experimental): 10ml twice a day for 4 Days.
  Interventions: Other: Hypertonic salt solution
- Essential oil mouthrinse (Active Comparator): 10ml twice a day for 4 Days.
  Interventions: Other: Essential oil
- Chlorhexidine Gluconate mouthrinse (Active Comparator): 10ml twice a day for 4 Days.
  Interventions: Other: Chlorhexidine Gluconate
- Distilled water (Placebo Comparator): 10ml twice a day for 4 Days.
  Interventions: Other: Distilled water

INTERVENTIONS:
Other: Licorice — Licorice, since years is known for its anti-inflammatory, antimicrobial, antiviral, antiprotozoal, antioxidative, hepatoprotective, cardioprotective, immunomodulatory and antitumour activity. Licorice can be beneficial for oral health. Glycyrrhizin, the sweet component of licorice root has antiplaque property. Pterocarpenes isolated from G. uralensis root extract exerts an antibacterial activity against Streptococcus mutans.
  Other Names: Glycyrrhiza
  Arms: Licorice extract mouthrinse
Other: Hypertonic salt solution — The antiseptic and bactericidal qualities of salt help in removing plaque which is a cause of gingivitis and caries. Warming water with a pinch of table salt can reduce or even be an alternative to anti-inflammatory drugs intra-orally. Its high osmolality reduces inflammation and can be microbicidal. Moreover, efficacy of luke warm hypertonic salt solution has shown antimicrobial, anti-inflammatory and immunomodulatory properties.
  Arms: Hypertonic salt solution
Other: Essential oil — Essential oils have a wide application in folk medicine, food flavoring and preservation as well as in fragrance industries. The antimicrobial properties of essential oils have been known for many centuries. In recent years, a large number of essential oils and their constituents have been investigated for their antimicrobial properties against some bacteria and fungi. Essential oils have the potential to be used as therapeutic agents for chronic gingivitis and periodontitis conditions that have both bacterial and inflammatory components.
  Arms: Essential oil mouthrinse
Other: Chlorhexidine Gluconate — Chlorhexidine is a symmetrical bisbiguanide synthetic antiseptic. It is available in three forms, digluconate, acetate and hydrochloride salts. Which have broad spectrum antimicrobial activity; it is effective against both Gram-positive and Gram-negative bacteria including aerobes and anaerobes, yeasts, fungi and lipid enveloped viruses. Chlorhexidine is considered to be the most effective plaque inhibitor against which other antiplaque agents are measured.
  Other Names: Chlorhexidine
  Arms: Chlorhexidine Gluconate mouthrinse
Other: Distilled water — Distilled water is commonly placebo in various research projects and it is also useful in as placebo treatment.
  Arms: Distilled water

SUMMARY:
Periodontal disease is a multifactorial disease caused by mainly bacterial, genetic, immunological, and environmental factors. Chronic periodontitis, one of the widely prevalent forms of periodontal disease, is characterized by loss of attachment apparatus of the tooth; it can lead to tooth loss. Many non surgical and surgical approaches have been adapted time and again to prevent, intercept, and to treat the various forms of chronic periodontitis. But, these treatment modalities are not approachable by all individuals, because of the various factors such as: low socioeconomic status, illiteracy, high cost of the treatment, no availability of easy and uncomplicated treatment nearby etc. Considering these factors, there are still a need of preventive, practical, and affordable treatment options specially for the population of underdeveloped and developing countries.

DETAILED DESCRIPTION:
Periodontal disease is a chronic inflammatory process accompanied by destruction of attachment apparatus of tooth and may lead to loss of teeth. It is a multifactorial disease, dental plaque being considered as primary etiologic factor in initiation and progression of disease. Control of periodontal disease by eliminating all pathogenic organisms of the microflora is, as yet, impossible but, it is theoretically an attractive aspect. Based on epidemiological studies there is a very strong correlation between the localization of dentogingival plaque and periodontal disease. Studies have clearly demonstrated that the ability to control the onset or progression of periodontal diseases is improved by regular plaque control practices. Although data shows that oral health can be improved through effective plaque control by mechanical means of cleaning but it fails to deliver optimal levels of oral health because the techniques are not being practiced consistently or thoroughly by all the individuals.

Over the past decade, various antimicrobial compounds have been investigated for their effectiveness to control plaque, but, chlorhexidine digluconate (CHX) is still being considered to be the most effective plaque inhibitor against which other antiplaque agents are measured. Chlorhexidine mouthwash is regarded as Gold standard mouthwash but has many local side effects: extrinsic brown staining of teeth and tongue, taste disturbance, enhanced supragingival calculus formation, desquamation of oral mucosa, and even liver damage in rats.

Cost effectiveness of chlorhexidine also matters especially in underdeveloped and developing countries where prevalence ratio of periodontal diseases are very high. The prevalence of gingivitis and periodontitis, along with their severity and rate of progression is found to vary worldwide; high in developing countries with approximately 80% prevalence in India.

Plant essential oils (EO) have the potential to be used as therapeutic agents for chronic gingivitis and periodontitis conditions that have both bacterial and inflammatory components. These are useful as their long term daily use has no adverse effects on the health of an individual. Also, these are more cost-effective and easily available as over-the-counter products.

It is need of the hour / high time to conduct the research work on various traditional oral hygiene practices / medicines to see their efficacy in the field of periodontics, as various uses of traditional medicine are still untouched & unexplored and few/no any such scientific documents are available, worldwide. And thus, attempts should be made to search for an alternative; Antiplaque, Plaque inhibitory, Anti gingivitis, Host modulating agent, and any other way acting on various levels of prevention of Gingival / Periodontal diseases by using traditional oral hygiene practices/ indigenous products/ homemade remedies/ medicines for maintenance of oral hygiene. Such research work may not only give an alternate antiplaque / plaque inhibitory, and anti-gingivitis agents but, at the same time may give different avenues in imparting treatment modalities on various levels of prevention of Gingival and Periodontal diseases. They may be more effective, more practical, less time consuming, and within the reach of each & every individual of the world in comparison to gold standard 'Chlorhexidine Gluconate Mouthrinse' and various other expensive therapeutic procedures.

Glycyrrhiza glabra (Licorice) (Family: Fabaceae) is one of the most important herbs and has been commonly utilised as ayurvedic medicine. It has been described as 'The grandfather of herbs' (Ody, 2000). In almost every Indian household you may find this herb chewed whenever someone's voice goes down. The earliest evidence regarding the use of licorice comes from the samples of licorice found in the tombs of Egyptian pharaohs, including those found in tomb of King Tut (1343 to 1325 BC). The main usage of licorice as a medicinal plant in European culture have been in the treatment of peptic ulcers and bronchial catarrhs. In Chinese herbal medicine, licorice is used as an expectorant, an analgesic, drug to treat asthma, drug to alleviate abscesses and abdominal pain. Licorice, since years is known for its anti-inflammatory, antimicrobial, antiviral, antiprotozoal, antioxidative, hepatoprotective, cardioprotective, immunomodulatory and antitumour activity.

There has been some indications that suggests licorice can be beneficial for oral health. One of the most important research has focussed on the benefits of water extract of licorice root for treatment of apthous ulcers. Glycyrrhizin, the sweet component of licorice root has antiplaque property. Pterocarpenes isolated from G. uralensis root extract exerts an antibacterial activity against Streptococcus mutans. So far, hardly any study has been conducted to see the antiplaque and antigingivitis effect of licorice as a traditional medicinal herb.

Life cannot exist without salt. Salt in various forms is being used since ages. 'Salt water' has been used by many cultures over countless generations to clean wounds and rinse mouths. Use of hot salt water rinsing is in practice to reduce the symptoms of pain in both gums and throat. It is also being routinely recommended following dental extraction, to keep food debris out of healing wounds and to reduce the incidence of alveolar osteitis. The antiseptic and bactericidal qualities of salt help in removing plaque which is a cause of gingivitis and caries. Warming water with a pinch of table salt can reduce or even be an alternative to anti-inflammatory drugs intra-orally. Its high osmolality reduces inflammation and can be microbicidal. Moreover, efficacy of luke warm hypertonic salt solution has shown antimicrobial, anti-inflammatory and immunomodulatory properties but its antiplaque efficacy is yet to be established with stabilised formula.

Above stated background have stimulated and encouraged us to conduct the study so, theinvestigators hypothesized the antiplaque efficacy of Licorice extract mouthrinse (LE) , 5% Hypertonic salt solution (HSS) as mouth rinses. Hence, the investigators planned this study titled "Evaluation of Antiplaque Efficacy of Licorice Extract Mouthrinse & 5% Hypertonic Salt Solution and their Comparison with Essential Oil & Chlorhexidine Mouthrinses-An Invitro & Invivo Study" with aforementioned aims and objectives.

ELIGIBILITY:
Inclusion Criteria:

* General/Medical

  1. Any race/ethnic group
  2. Aged - 18-30 years
  3. Male or female
  4. No acute or chronic systemic conditions (see exclusion criteria below)
  5. No medications/medication history that can interfere with the study (see exclusion criteria below)
  6. Non-smoker, Non-alcoholic
  7. Who was ready to comply with study procedures
  8. Who was available for the duration of the study
  9. Who were ready to provide signed informed consent Oral/Periodontal

  <!-- -->

  1. Dentate with at least 14 natural teeth, excluding third molars, that can be evaluated periodontally.
  2. Patients with Healthy periodontium and/or Mild Gingivitis.
  3. No acute oral diseases (mucosal lesions), oral infections, need for immediate dental/periodontal care (e.g., NUG).

Exclusion Criteria:

* General/Medical A) Any known systemic disease which has effects on periodontium such as diabetes, cardiovascular, cancer etc.

B) Volunteers on anti-inflammatory, antibiotics, steroids, cytotoxic, and perioceutics, since 03 months.

C) Volunteers who are known allergic to any substance. D) Pregnant and lactating mothers. E) Volunteers who had dental caries. F) Tobacco users (smoke and smokeless) and Alcoholics. G) Volunteers wearing any form of intraoral prosthesis or appliance. Oral/Periodontal

1. <14 teeth that can be periodontally evaluated (excluding 3rd molars)
2. Dental volunteers with compromised periodontal status/ any sign of moderate or severe gingivitis and periodontitis.
3. Acute oral infections.
4. Oral wounds, including recent extractions.
5. Patients with removable or fixed orthodontic appliances

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-06-10 (Actual)

PRIMARY OUTCOMES:
Modified Plaque Index | After 4 days
  Modified Plaque Index (Turesky, Gilmore, Glickman modification of Quigely Hein Index, 1970) after disclosing the teeth with two tone solution the PI was recorded. Facial and lingual aspects were scored with PI. Scoring was as follows: 0 - No plaque/debris 1 - Separate flecks of plaque at the cervical margin of the tooth. 2 - A thin continuous band of plaque (up to 1mm) at the cervical margin of the tooth. 3 - A band of plaque wider than 1 mm but covering less than one third of the crown of the tooth 4 - plaque covering at least one third but less than two thirds of the crown of the tooth. 5 - Plaque covering two third or more of the crown of the tooth. Modified Plaque Index = Total score / no. of surfaces examined.

OTHER OUTCOMES:
Minimum inhibitory concentration | 72 hours
  Minimum inhibitory concentration (MIC) is the lowest concentration of an antimicrobial (like an antifungal, antibiotic or bacteriostatic) drug that will inhibit the visible growth of a microorganism after overnight incubation). Tested against following periopathogens: Porphyromona sgingivalis, Prevotella intermedia, fusobacteriumnucleatum, Aggregatibacter actinomycetemcomitans, Capnocytophaga, Tannerella forsythia, Pseudomonas aeruginosa, Streptococcus mutans, E. faecalis, and Candida.
Minimum bactericidal concentration | 72 hours
  Minimum bactericidal concentration (MBC) is the lowest concentration of an antibacterial agent required to kill a particular bacterium. It can be determined from broth dilution minimum inhibitory concentration (MIC) tests by sub culturing to agar plates that do not contain the test agent. Tested against following periopathogens: Porphyromonas gingivalis, Prevotella intermedia, fusobacterium nucleatum, Aggregatibacter actinomycetemcomitans, Capnocytophaga, Tannerella forsythia, Pseudomonas aeruginosa, Streptococcus mutans, E. faecalis, and Candida.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Subhash Garg, Study Chair — Govt. College of Dentistry Indore, M.P. India,Indore, M.P, India, 452001

IPD SHARING:
Plan to Share IPD: Undecided